CLINICAL TRIAL: NCT05658120
Title: Risk Factors and Postoperative Complications of Reperfusion Syndrome and Vasoplegic Syndrome in Patients With Vasoactive Support During Liver Transplant Surgery
Brief Title: Reperfusion Syndrome and Vasoplegic Syndrome in Liver Transplant Surgery
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)460/2017
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-12

CONDITIONS: Postperfusion Syndrome
Keywords: postreperfusion syndrome; vasoplegic syndrome
MeSH Terms: conditions — Vasoplegia | interventions — Norepinephrine; Epinephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: noradrenaline/adrenaline — norepinephrine adrenaline in patients with Swan-Ganz catheter monitoring during liver transplantation
  Other Names: Swan-Ganz catheter monitoring

SUMMARY:
The incidence of postreperfusion syndrome (PRS) and vasoplegic syndrome (VS) is unknown, and occasionally can be confused since these syndromes share some hemodynamic characteristics. In these cases, monitoring with Swan Ganz catheter may be useful to make the differential diagnosis. The main outcome was to analyze reperfusion syndrome and vasoplegic syndrome in patients receiving vasoactive support during liver transplant surgery, in terms of incidence, risk factors and postoperative complications.

DETAILED DESCRIPTION:
Introduction:

At the time of the liver reperfusion, many inflammatory mediators coming from the liver graft to the systemic circulation produce a sudden load of cold and acidotic blood. At this stage of graft revascularization, it has been seen an increase of pulmonary vascular resistance index (PVRI) and pulmonary arterial pressure (PAP) and a reduction in systemic vascular resistance index (SVR), heart rate (HR), cardiac index (CI) and arterial blood pressure (ABP).

In this context, some patients suffer postreperfusion syndrome (PRS). This syndrome was first defined by Aggarwal et al as a decrease in the MAP greater than 30% of at least one minute duration and during the five minutes following the portal unclamping and was associated with several preoperative risk factors and postoperative complications. The variety of the risk factors presented in previous studies suggest that the PRS occurs in an unpredictable manner. These risk factors were described related to the organ of the donor; related to the recipient of the liver graft, and related to the surgical technique. The incidence varies largely among the considered studies, ranging from 12% to 77% and it can respond not only to preoperative and intraoperative factors associated with anesthetic-surgical practice, but also to the different criteria for definition of PRS as well as to the administration of vasoactive drugs to prevent or treat it.

On the other hand, the incidence of vasoplegic syndrome (VS) is not described and could be confused with PRS We studied the patients who received vasoactive support during liver transplant surgery and presented PRS considering the Aggarwal et al. definition, and VS considering the Ozal et al. criteria.

Methods:

Design: Retrospective observational study. Inclusion criteria: Patients undergoing liver transplantation who received vasoactive support and monitored with Swan Ganz catheter Exclusion criteria: liver transplantation for acute liver failure, combined liver and kidney transplantation, renal dysfunction (glomerular filtration <60), moderate/severe vascular and valvular heart disease, moderate/severe hepatopulmonary syndrome, moderate/severe portopulmonary syndrome, and re-transplantation

* Study outcomes The primary objective of our study was to determine the incidence and risk factors of PRS and VS in norepinephrine/adrenaline patients according to the Aggarwal and Ozal criteria respectively. The second objective is to determine the postoperative complications.
* Data collection Preoperative variables related to recipient and donor were analyzed. Intraoperative variables were recorded at each stage of the surgery: pulmonary capillary wedge pressure (PCWP), mean pulmonary arterial pressure (mPAP), MAP, heart rate (HR), cardiac index (CI), systemic vascular resistance index (SVRI), central venous pressure (CVP), bleeding, need for transfusions, doses of vasoconstrictors, global requirements for bicarbonate and calcium chloride, presence of malignant arrhythmias (fibrilation, flutter, ventricular tachycardia) or ischemic electrocardiographic abnormalities. The times of each surgical phase, duration of cold ischemia and the weights of the liver (donor/recipient) were recorded too. Postoperative data collected included: graft rejection, a second surgery after liver transplant, the need for re-transplantation, renal dysfunction (glomerular filtration <60), hospital stay, days of hospitalization and survival.

All items that could be used to identify the patient (clinical record ID number or name) were removed to protect personal data.

-Measurement of hemodynamic data The hemodynamic parameters (MAP, HR, SVR, CVP, CI, PCWP and mPAP) of each stage of the liver transplant surgery (dissection phase, anhepatic phase prior to unclamping of the IVC, at 1 and 5 min after graft reperfusion, and in the neohepatic phase after completion of the vascular anastomosis) were collected.

The PRS criteria were decrease in the mean arterial pressure ≥ 30% mmHg during the first 5 minutes after unclamping of the IPV, decrease in CI and SVR respect to baseline (anhepatic phase), and increase of the PCWP, CVP and mPAP respect to baseline.

Association between PRS and preoperative, intraoperative, and postoperative variables were analyzed and compared between the two groups (for PRS + and PRS - groups).

ELIGIBILITY:
Inclusion Criteria: Consecutive patients ≥ 18 years-old, who underwent liver transplant surgery, monitored with Swan-Ganz catheter, with norepinephrine/adrenaline support during transplant surgery

Exclusion Criteria:

Acute liver failure, combined liver/kidney transplantation, re-transplantation, living-donor related transplantation, moderate to severe vascular and valvular heart disease, chronic kidney disease (serum creatinine > 1.5), moderate and sever hepato-pulmonary syndrome, moderate and sever porto-pulmonary syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients ≥ 18 years-old, who underwent liver transplant surgery, monitored with Swan-Ganz catheter, with norepinephrine/adrenaline support during transplant surgery
Sampling Method: Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-02-18 (Actual)

PRIMARY OUTCOMES:
incidence of PRS and VS | in the first 5 min after vascular unclamping
  Incidence of PRS and VS in patients undergoing liver transplantation

SECONDARY OUTCOMES:
postoperative complications | 3 months
  Determie the postoperative complications in patients with PRS and VS

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d´Hebron Research Institute VHIR, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
there is no plan

REFERENCES:
- [Background] Ozal E, Kuralay E, Yildirim V, Kilic S, Bolcal C, Kucukarslan N, Gunay C, Demirkilic U, Tatar H. Preoperative methylene blue administration in patients at high risk for vasoplegic syndrome during cardiac surgery. Ann Thorac Surg. 2005 May;79(5):1615-9. doi: 10.1016/j.athoracsur.2004.10.038. PMID 15854942
- [Result] Aggarwal S, Kang Y, Freeman JA, Fortunato FL, Pinsky MR. Postreperfusion syndrome: cardiovascular collapse following hepatic reperfusion during liver transplantation. Transplant Proc. 1987 Aug;19(4 Suppl 3):54-5. No abstract available. PMID 3303534